CLINICAL TRIAL: NCT05590078
Title: Evaluation of Interest of LUMEEN Virtual Reality Headset to Reduce Preoperative Anxiety in AMBulatory Surgery
Acronym: AMBLUMEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0102
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Anxiety
Keywords: Virtual reality; preoperative anxiety; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): General routine care. This group will undergo to ambulatory surgery without preoperative virtual reality session. Will be applied the usual treatment to reduce preoperative anxiety.
  Interventions: Other: State Trait Anxiety Inventory; Other: Perioperative care satisfaction score
- Virtual reality group (Experimental): Virtual Reality. This group will undergo to 20 min virtual reality before ambulatory surgery. In addition to virtual reality session, will be applied the usual treatment to reduce preoperative anxiety, after virtual reality, if necessary.
  Interventions: Device: Virtual reality session; Other: State Trait Anxiety Inventory; Other: Virtual Reality Satisfaction Score; Other: Perioperative care satisfaction score

INTERVENTIONS:
Device: Virtual reality session — The 20-minute virtual reality session, in the outpatient department before surgery, immerses the patient in calm environments combined with music therapy and breathing exercises to relax and reduce anxiety.
  Arms: Virtual reality group
Other: State Trait Anxiety Inventory — The State Trait Anxiety Inventory (State anxiety) is a questionnaire given to adults that shows how strong a person's feelings of anxiety are "right now, just now". The score is measured on arrival in the outpatient department and just before going into the intervention room (= after the virtual reality session for the experimental group)
Other: Virtual Reality Satisfaction Score — Likert scale satisfaction questionnaire to collect the patients' satisfaction regarding virtual reality session
  Arms: Virtual reality group
Other: Perioperative care satisfaction score — Likert scale satisfaction questionnaire to collect the patients' satisfaction regarding perioperative care

SUMMARY:
This study evaluate the interest of Virtual Reality to reduce the preoperative anxiety in patients who undergo to ambulatory surgery. Half of the patients will received the virtual reality program, and the other half will received de common treatment.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II (classification of the American Society of Anesthesiologists).
* Ambulatory surgery scheduled
* Score STAI YA > 45
* Affiliated to a social security
* Understanding the study and signing the informed consent

Exclusion Criteria:

* Contraindications for Midazolam
* Patients with disorders not compatible with virtual reality: severe cognitive or psychiatric disorders, blindness, claustrophobia, epilepsy
* Patient with a pacemaker of others implantable medical devices
* patient with burns or wounds on the upper face or scalp
* Visual hallucinations
* Contagious disease by air or indirect contact
* Person unable to express their consent
* Minor patient or patient under curatorship or guardianship
* patient participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Change of Anxiety | D0 : baseline and right before going to surgery
  Measured by State-Trait Anxiety Inventory (STAI YA) . The scale includes twenty items.. Each question is assigned 1 to 4 points, giving a score of 20 (low anxiety) to 80 points (high anxiety)

SECONDARY OUTCOMES:
Number of milligrams of midazolam administered | D0 (before surgery)
  Comparison of midazolam premedication to reduce preoperative anxiety between control group and virtual reality group.
Percentage of patients with intraoperative remifentanil required | D0 (during surgery)
  Comparison in term of Number of case where the utilisation of remifentanil was necessary in peroperative between control group and virtual reality group.
Pain score | D0 (after surgery)
  Pain assessment with numerical scale from 0 (low) to 10(high)
Morphine dose used | D0 (after surgery in recovery room)
  Comparison of morphine dose used in recovery room between control group and virtual reality group
Perioperative care satisfaction score | through study completion, 1 day
  Likert scale satisfaction questionnaire to collect the patients' satisfaction regarding perioperative care. 5 answer possible :Very satisfied - satisfied- Neither satisfied nor unsatisfied- Unsatisfied - Very unsatisfied
Nature and severity of adverse events | through study completion, 1 day
  Comparison of adverse event during hospitalization between control group and virtual reality group
Adverse events related to the virtual reality session | through study completion, 1 day
  Nature and severity of adverse events related to the virtual reality session
Virtual Reality Satisfaction Score | through study completion, 1 day
  Likert scale satisfaction questionnaire to collect the patients' satisfaction regarding virtual reality session. 5 items scored from 0 (low) to 10 (high)
Experience of the caregiver | D0 (before surgery)
  Experience of the caregiver concerning the implementation of virtual reality in the outpatient department before surgery . 2 items scored from 0 (low) to 10 (high)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud FRIGGERI, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No